CLINICAL TRIAL: NCT01939093
Title: Therapeutic Effect Between Quetiapine and Haloperidol on the Treatment of Methamphetamine - Induced Psychosis
Brief Title: Therapeutic Effect of Quetiapine on Methamphetamine-Induced Psychosis
Acronym: MAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Thanyarak Institute (Unknown); National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Rasmon Kalayasiri, Assistant Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRCT-53069
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Methamphetamine-induced Psychosis
Keywords: Quetiapine; Haloperidol; Methamphetamine; Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Diazepam; Cinnarizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine (Experimental): Quetiapine 100 mg per day is taken orally once a day for four weeks. The dose is increased every 5 days until no psychotic symptom is observed.
  Interventions: Drug: Diazepam; Dietary Supplement: Vitamin B1-6-12; Drug: Stugeron
- Haloperidol (Active Comparator): Haloperidol 2 mg per day is taken orally once a day for four weeks. The dose is increased every 5 days until no psychotic symptom is observed.
  Interventions: Drug: Diazepam; Dietary Supplement: Vitamin B1-6-12; Drug: Stugeron

INTERVENTIONS:
Drug: Diazepam — If subjects had aggressive or violent symptoms and immediate symptom control was needed, 10 mg of diazepam (intravenous injection) every 4 hours is allowed for symptom control.
Dietary Supplement: Vitamin B1-6-12 — All subjects will be given the Institute's medication regimen, including vitamin B1-6-12 1 tablet three times a day after meals during the whole study period.
Drug: Stugeron — All subjects will be given the Institute's medication regimen, including stugeron 1 tablet three times a day after meals during the whole study period.

SUMMARY:
The aims of this study are to compare the antipsychotic and adverse events of quetiapine, an atypical antipsychotic drug, to haloperidol, a standard treatment for primary psychotic disorder, in individuals with MAP.

DETAILED DESCRIPTION:
Eighty individuals with MAP will be randomly assigned into two treatment groups, i.e. treatment with quetiapine and haloperidol. The quetiapine group will receive quetiapine at least 100 mg per day and the haloperidol group will receive haloperidol at least 2 mg per day orally once a day for four weeks. The doses will be increased every 5 days until no psychotic symptom is observed from the Positive and Negative Syndrome Scale. Common antipsychotic adverse events will be checked and documented daily.

ELIGIBILITY:
Inclusion Criteria:

* Having a psychotic episode with current use of methamphetamine
* Positive urine toxicology test for methamphetamine on the first day of hospitalization

Exclusion Criteria:

* Using other illegal substances
* Having a history of primary psychotic disorders or using antipsychotic agents
* Having a chronic medical disease, e.g. essential hypertension, diabetes, epilepsy, stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | Every day in Week 1.
Positive and Negative Syndrome Scale | Every two days in Week 2 and 3.

SECONDARY OUTCOMES:
Antipsychotic Adverse Event Form | Every day for three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Viroj Verachai, M.D., Principal Investigator — Thanyarak Institute on Drug Abuse
Locations (1):
- Thanyarak Institute on Drug Abuse, Pathum Thani, Changwat Pathum Thani, Thailand